CLINICAL TRIAL: NCT06151964
Title: A Phase I/II, Randomised, Single-blind, Placebo-controlled, Multiple-ascending-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AZD9550 Monotherapy and Co-administration of AZD9550 and AZD6234 in Participants Living With Obesity and Overweight With or Without Type 2 Diabetes Mellitus
Brief Title: A Trial to Learn How Safe AZD9550 Monotherapy and Combined With AZD6234 is in People With or Without Type 2 Diabetes Who Are Living With Obesity and Overweight
Acronym: CONTEMPO
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D8460C00002; 2023-504215-32-00 (Registry Identifier: EU CT)
Record Dates: First submitted 2023-09-22; First posted 2023-11-30 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Overweight and Obesity
Keywords: AZD9550; AZD6234; Non-alcoholic Fatty Liver Disease; Non-alcoholic Steatohepatitis; Overweight; Obese; Obesity; Diabetes Mellitus, Type 2; Liver Glycogen; Adipose Tissue; Glucose; 3-Hydroxybutyric Acid; Subcutaneous Fat; Liver fat; Magnetic Resonance Imaging; Magnetic Resonance Spectroscopy; Weight Loss; Mixed Meal Tolerance Test
MeSH Terms: conditions — Overweight; Obesity; Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2; Fatty Liver; Weight Loss

STUDY DESIGN:
Intervention Model Description: The study will randomise approx. 120 participants and is devided in 5 parts (Part D conducted only in Japan):
  A: Approx. 45 participants will be screened to achieve 16 randomised. The study duration approx. 103 days.
  B: Approx. 90 participants will be screened to achieve 30 randomised. The study duration approx. 110 days.
  C: Approx. 90 participants will be screened to achieve 30 randomised. The study duration approx. 249 days.
  D: Approx. 35 participants will be screened to achieve 12 randomised. The study duration approx. 249 days.
  E: Approx. 80 participants will be screened to achieve approx. 28 randomised. The study duration approx. 249 days.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This study is single-blind with regard to treatment (AZD9550 monotherapy, co-administered AZD9550 and AZD6234, or placebo). This means that the participant, investigator, Study Monitor, and the clinical unit staff will remain blinded during each part of the study and the randomisation code will only be available at each predefined decision point before the SRC meeting in order to review the data unblinded, if necessary. The sponsor will be unblinded throughout the study.
  AZD9550, AZD6234, and placebos will as far as possible be matched for appearance and volume. Participants randomised to placebo will receive the same volume of injection (SC cohorts) as participants on active treatment. In Part E, the number of injections per dosing occasion (ie, 2) will be the same in all treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Part A: AZD9550 (Experimental): Multiple repeat doses of AZD9550 given as 4 once weekly SC doses for 4 weeks to 2 sequential cohorts in overweight/obese participants with or without T2DM, evaluating 2 low dose levels of AZD9550
  Interventions: Drug: AZD9550
- Part B: AZD9550 (Experimental): Once weekly up-titration over 5 doses of AZD9550 in overweight/obese participants with or without T2DM
  Interventions: Drug: AZD9550
- Part C: AZD9550 (Experimental): Bi-weekly/monthly up-titration of AZD9550 for 24 weeks in overweight/obese participants with or without T2DM.
  Interventions: Drug: AZD9550
- Part D: AZD9550 (Experimental): Bi-weekly/monthly up-titration of AZD9550 for 24 weeks in overweight/obese Japanese participants with T2DM.
  Interventions: Drug: AZD9550
- Part A: placebo (Experimental): Multiple repeat doses of placebo given as 4 once weekly SC doses for 4 weeks to 2 sequential cohorts in overweight/obese participants with or without T2DM, evaluating 2 low dose levels of AZD9550
  Interventions: Drug: Placebo
- Part B: placebo (Experimental): Once weekly administration of placebo over 5 doses, volume matched to the active treatment being up-titrated, in overweight/obese participants with or without T2DM
  Interventions: Drug: Placebo
- Part C: placebo (Experimental): Bi-weekly/monthly administration of placebo - volume matched to the active treatment being up-titrated - for 24 weeks in overweight/obese participants with or without T2DM.
  Interventions: Drug: Placebo
- Part D: placebo (Experimental): Bi-weekly/monthly administration of placebo - volume matched to the active treatment being up-titrated - 24 weeks in overweight/obese Japanese participants with T2DM.
  Interventions: Drug: Placebo
- Part E: AZD9550 and AZD6234 (Experimental): Bi-weekly/monthly up-titration of AZD9550 and AZD6234 for 24 weeks in overweight/obese participants with T2DM.
  Interventions: Drug: AZD9550 and AZD6234
- Part E: Placebo (Experimental): Bi-weekly/monthly administration of placebo - volume matched to the active treatments being up-titrated - 24 weeks inoverweight/obese participants with T2DM.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD9550 — Part A: A constant dose Part B: Doses of AZD9550 that increase each week Part C: Doses of AZD9550 that increase every 2 weeks, then every 4 weeks Part D: Doses of AZD9550 that increase every 2 weeks, then every 4 weeks
  Arms: Part A: AZD9550; Part B: AZD9550; Part C: AZD9550; Part D: AZD9550
Drug: Placebo — Matching administration volumes for SC injection
  Arms: Part A: placebo; Part B: placebo; Part C: placebo; Part D: placebo; Part E: Placebo
Drug: AZD9550 and AZD6234 — Part E: Doses of AZD9550 and AZD6234 that increase every 2 weeks, then every 4 weeks
  Arms: Part E: AZD9550 and AZD6234

SUMMARY:
AZD9550, previously being developed for the treatment NASH, is a dual GCG and GLP-1 receptor agonist. AZD9550 is now being developed in combination with AZD6234, a SARA, for the treatment of overweight and obesity and its associated co-morbidities. Co-administration of AZD9550 and AZD6234 is currently being evaluated in participants living with obesity and overweight without T2DM in an ongoing Phase 2b study.

The purpose of this study is to investigate the safety, tolerability, and effects of increasing doses of AZD9550 monotherapy in overweight and obese participants aged 18 through 65 years living with or without T2DM, and to investigate how AZD9550 is absorbed, distributed, and eliminated from the body (Parts A-D).

In addition, the study will investigate the safety and tolerability of co-administration of AZD9550 and AZD6234 in participants living with T2DM with obesity or overweight aged 18 through 75 years (Part E).

DETAILED DESCRIPTION:
This Phase I/II, randomised, single-blind, placebo-controlled, MAD study will assess the safety and tolerability of AZD9550 monotherapy and co-administration of AZD9550 and AZD6234 and will characterise the PK and PD of AZD9550 monotherapy and co-administration of AZD9550 and AZD6234 following SC administration to overweight and obese participants living with or without T2DM. Inclusion of participants receiving placebo is appropriate for benchmarking the safety and tolerability of AZD9550 and co-administration of AZD9550 and AZD6234. A randomised and single-blind study design has been chosen to minimise bias and includes a placebo to facilitate identification of effects related to the administration of the study intervention rather than the study procedures or situation.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 through 65 years (Parts A-D) or 75 years (Part E) at the time of screening.
2. Parts A, B, C only: Participants with or without T2DM. If participants have a diagnosis of T2DM, the glucose control managed with diabetes diet and in addition to metformin treatment no more than two treatment options (with a stable dose 3 months prior to screening).

   Part D only: Participants who are diagnosed with T2DM, have inadequate glycaemic control with diet and exercise. Participants who are prescribed an oral anti-diabetic agent such as metformin, a DPP IV inhibitor, sulphonylurea, glinides, alphaglucosidase inhibitors, and an SGLT2 inhibitor may be eligible to enter the study following a washout of 4-weeks or 5-half lives (whichever is longer) washout period.

   Part E only: Participants are eligible to be included in the Part E only if they meet all of the following criteria at screening:
   1. Diagnosed with T2DM.
   2. Are treated with diet and exercise only, or any combination of OAD with stable doses in the 3 months prior to dosing.
   3. Participants prescribed a DPP IV inhibitor or a GLP-1RA-containing medicine, alone or in combination with other OADs, may be eligible to enter the study if they have not been treated with any of these drugs for at least 35 days or 5 drug half-lives (whichever is longer) prior to randomisation.
3. Participants with a screening HbA1c value within the target range of

   • ≥ 42 to ≤ 86 mmol/mol (6% to 10%).
4. Body mass index from ≥27 (≥25 in Part D) to ≤39.9 kg/m2 (inclusive) (Part A-D) or ≥ 27 kg/m2 (Part E).
5. Contraceptive use by males or females should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
6. Written informed consent and any locally required authorization (eg, European Union Data Privacy Directive) obtained from the participant prior to performing any protocol-related procedures, including screening evaluations
7. Ability to complete and meet all eligibility requirements for randomisation within 60 days after signing the ICF.
8. Venous access suitable for multiple cannulations.
9. Willing and able to self-administer weekly SC injections (Parts C, D and E only).

Exclusion Criteria:

1. Participants with T2DM treated with insulin.
2. Participants with T2DM treated with more than 3 anti-diabetic therapies (Parts A-D only).
3. Participants with or without T2DM treated with a GLP-1RA or GLP-1RA/GIPRA within 3 months of screening (Parts A to D only) or within 35 days of randomisation or five half-lives (whichever is shorter) of dosing (Part E only).
4. History of any clinically important disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
5. Serum calcitonin suggestive of thyroid C-cell hyperplasia (calcitonin level > 50 ng/L), medullary thyroid carcinoma, or history or family history of multiple endocrine neoplasia at screening.
6. History or presence of GI, renal, or hepatic disease (with the exception of Gilbert's syndrome), or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs, as judged by the investigator.
7. History of cancer within the last 10 years, with the exception of non-melanoma skin cancer.
8. Any clinically important illness (apart from T2DM), as judged by the investigator.
9. Any medical/surgical procedure, or trauma within 4 weeks prior to screening, at the discretion of the investigator.
10. Symptoms of insulinopenia or poor blood glucose control (eg, significant thirst, nocturia, polyuria, polydipsia, or weight loss).
11. Positive hepatitis B or hepatitis C virus serology at screening.
12. Positive human immunodeficiency virus test at screening or participant taking antiretroviral medications as determined by medical history or participant's verbal report.
13. At screening blood tests, any of the following:

    * AST ≥ 1.5 × ULN
    * ALT ≥ 1.5 × ULN
    * TBL ≥ 1.5 × ULN (with the exception of Gilbert's syndrome)
    * Haemoglobin below the lower limit of the normal range or any other clinically significant haematological abnormality as judged by the investigator.
    * Total serum calcium, albumin-corrected calcium or ionised calcium < LLN at screening (Part E).
14. Impaired renal function defined as estimated glomerular filtration rate (eGFR) ≤ 60 mL/minute/1.73m2 as defined by Chronic Kidney Disease Epidemiology Collaboration (2021) (Part A to D); or ≤ 45 mL/minute/1.73 m2 (Part E).
15. Any clinically important abnormalities in clinical chemistry, haematology, coagulation, or urinalysis results other than those specifically described as exclusion criteria herein, as judged by the investigator.
16. Significant late diabetic complications (macroangiopathy with symptoms of congestive heart disease or peripheral arterial disease, microangiopathy with symptoms of neuropathy, gastroparesis, retinopathy requiring treatment, nephropathy) detected in laboratory results or in clinical history/documentation as judged by the investigator.
17. Abnormal vital signs, after 10 minutes of supine rest, defined as any of the following:

    * Systolic BP < 90 mmHg or ≥ 150 mmHg
    * Diastolic BP < 50 mmHg or ≥ 90 mmHg
    * HR < 50 or > 85 bpm at resting state
    * Participants may be re-tested for the vital signs criteria only once if, in the investigator's judgement, they are not representative of the participant.
18. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG and any abnormalities in the 12-lead ECG that, as considered by the investigator, may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology or left ventricular hypertrophy.
19. Participants with implantable cardiac defibrillator or a permanent pacemaker, and participants with symptomatic tachy- or brady-arrhythmias.
20. Participants with unstable angina pectoris or stable angina pectoris classified higher than Canadian Cardiovascular Society class II or an acute coronary syndrome/acute myocardial infarction or coronary intervention with percutaneous coronary intervention or coronary artery bypass grafting or stroke within 6 months.
21. In Parts A-D: History of hospitalisation caused by heart failure or a diagnosis of heart failure. In Part E, severe congestive heart failure (New York Heart Association Class III or IV) or recent (< 6 months) hospitalisation due to heart failure.
22. Known or suspected history of drug abuse within the past 3 years as judged by the investigator (Parts A-E) and or a positive screen for drugs of abuse at screening (Parts A-D only).
23. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity as judged by the investigator.
24. Whole blood or red blood cell donation, or any blood loss > 500 mL (or > 400 mL in Part D) during the 3 months prior to screening.
25. History of psychosis or bipolar disorder.
26. History of major depressive disorder within the 2 years prior to screening or depression, where the participant is deemed to be clinically unstable as judged by the investigator.
27. Previous hospitalisation for any psychiatric reason.
28. PHQ-9 score ≥ 15 within the 2 years prior to screening or at screening.
29. Received another new chemical entity (defined as a compound that has not been approved for marketing), or has participated in any other clinical study that included drug treatment within at least 30 days or 5 half-lives prior to the first administration of study intervention in this study (whichever is longer). The period of exclusion to begin 30 days or 5 halflives of IMP after the final dose, or after the last visit, whichever is longest. Participants consented and screened, but not randomised into this study or a previous Phase 1 study, are not excluded.
30. History of lactic acidosis
31. Use of any of the following medicinal products:

    * Use of systemic corticosteroids within 28 days prior to screening.
    * Use of compounds known to prolong the QTc interval.
    * Use of any herbal preparations or medicinal products licensed for control of body weight or appetite within 3 months prior to screening.
32. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of study intervention.
33. Received another new chemical entity (defined as a compound that has not been approved for marketing), or has participated in any other clinical study that included drug treatment within at least 30 days or 5 half-lives prior to the first administration of study intervention in this study (whichever is longer). The period of exclusion to begin 30 days or 5 half-lives of IMP after the final dose, or after the last visit, whichever is longest. Participants consented and screened, but not randomised into this study or previous AZD9550, AZD6234, or AZD9550/AZD6234 combination studies, are not excluded from Part E.
34. Previous enrolment or randomisation in the present study.
35. Concurrent participation in another study of any kind is prohibited.
36. Ongoing weight loss diet (hypocaloric diet) or use of weight loss agents, unless the diet or treatment has been stopped at least 3 months prior to screening and the participant has had a stable body weight (± 5%) during the 3 months prior to screening.
37. Participants who are vegans, ones with medical dietary restrictions, or participants who are willingly conducting any diet likely to increase ketone levels (Atkins or any similar diet based on increased protein consummation or low carbohydrate content) (Part A-D only).
38. Excessive intake of caffeine-containing drinks or food (eg, coffee, tea, Coca-Cola/Pepsi or similar drink type, chocolate) as judged by the investigator (Part A-D only).
39. Current smokers or those who have smoked or used nicotine products (including e-cigarettes) within the previous 3 months prior to screening (Part A-D only).
40. Participants who cannot communicate reliably with the investigator or vulnerable participants (eg, kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order).
41. The participant is an employee, or close relative of an employee, of AstraZeneca, the CRO, or the study site, regardless of the employee's role.
42. Judgement by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.
43. Contra-indication to MRI: such as participants with pacemakers, metallic cardiac valves, magnetic material such as surgical clips, implanted electronic infusion pumps or other conditions that would preclude proximity to a strong magnetic field; participants with history of extreme claustrophobia or participant cannot fit inside the MRI scanner cavity (Parts B and C only).
44. Serum triglyceride concentrations > 500 mg/dL (5.6 mmol/L) at screening or any other metabolic condition judged by the investigator as likely to precipitate acute pancreatitis (Part E only).
45. History of use of marijuana or THC-containing products within 3 months prior to screening or unwillingness to abstain from marijuana or THC-containing products use during the study (Part E only).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2027-03-17 (Estimated); Study Completion 2027-03-17 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of participants with any AE, SAEs, AEs leading to discontinuation of study intervention, AEs with outcome of death, and AEs leading to withdrawal from study. | Day - 35 to Day 205
  Applicable for Parts A, B, C, D, E.
Number and percentage of participants with clinically significant changes from baseline in Vital Sign Parameters. | Day - 35 to Day 205
  Applicable for Parts A, B, C, D, E.
Number and percentage of participants with clinically significant changes in ECG parameters. | Day - 35 to Day 205
  Applicable for Parts A, B, C, D, E.
Number and percentage of participants with clinically significant changes from baseline in Clinical Laboratory Parameters | Day - 35 to Day 205
  Applicable for Parts A, B, C, D, E.
Area Under Concentration-Time Curve of AZD9550 following repeat weekly SC doses | Day 1 to Day 65
  * AUC from 0 to the time of the last measured concentration (AUClast) at first dose and last dose
  * AUC over a dosing interval (AUCtau) at first dose and last dose.
  Applicable for Part A.
Maximum observed concentration of AZD9550 following repeat weekly SC doses | Day 1 to Day 65
  • Cmax at first dose and last dose
  Applicable for Part A.
Half life associated with terminal phase elimination rate constant of AZD9550 following repeat weekly SC doses | Day 1 to Day 65
  • t1/2λz at first dose and last dose
  Applicable for Part A.
Time to maximum observed concentration of AZD9550 following repeat weekly SC doses | Day 1 to Day 65
  • tmax at first dose and last dose
  Applicable for Part A.
Apparent oral clearance of AZD9550 following repeat weekly SC doses | Day 1 to Day 65
  • CL/F at first dose and last dose
  Applicable for Part A.
Apparent volume of distribution of AZD9550 following repeat weekly SC doses | Day 1 to Day 65
  • Vz/F at first dose and last dose
  Applicable for Part A.
Ratio for AUC of AZD9550 following repeat weekly SC doses | Day 1 to Day 65
  • Rac AUCtau at last dose
  Applicable for Part A.
Ratio for Cmax of AZD9550 following repeat weekly SC doses | Day 1 to Day 65
  • Rac Cmax at last dose
  Applicable for Part A.

SECONDARY OUTCOMES:
PD effect of AZD9550 on fasting glucose compared to placebo | From baseline to Week 4
  • Absolute change in fasting glucose
  Applicable for Part A.
PD effect of AZD9550 on fasting lipid profile compared to placebo | From baseline to Week 4
  • Absolute and percentage change in total cholesterol, high-density lipoprotein, low-density lipoprotein, triglycerides, and BHB
  Applicable for Part A.
Absolute and percentage change in body weight from baseline | From baseline to Week 4
  Applicable for Part A.
Incidence of anti-AZD9550 antibodies | From Day 1 to Day 65
  • Incidence of ADA to AZD9550
  Applicable for Part A.
Absolute change in percentage body fat from baseline | From baseline to Week 4
  Applicable for Part A.
PD effect of AZD9550 on fasting glucose compared to placebo | From baseline to Week 5
  • Absolute change in fasting glucose
  Applicable for Part B.
PD effect of AZD9550 on fasting lipid profile compared to placebo | From baseline to Week 5
  • Absolute and percentage change in total cholesterol, high-density lipoprotein, low-density lipoprotein, triglyceride, and BHB
  Applicable for Part B.
Effect of AZD9550 on hepatic fat fraction versus placebo at Week 5 | From baseline to Week 5
  * Change in hepatic fat fraction as measured by MRI-PDFF
  * Percent change in hepatic fat fraction as measured by MRI-PDFF
  Applicable for Part B.
PD effect of AZD9550 on glucose metabolism following an MMTT compared to placebo | From baseline to Week 5
  * Percent change in glucose AUC(0-4h) measured by MMTT
  * Percent change in insulin AUC(0-4h) measured by MMTT
  * Percent change in c-peptide AUC(0-4h) measured by MMTT
  Applicable for Part B.
Area Under concentration-time Curve of AZD9550 following repeat weekly SC doses | Day 1 to Day 72
  * AUC from 0 to the time of the last measured concentration (AUClast) at the last dose
  * AUC over a dosing interval (AUCtau) at first dose and last dose
  Applicable for Part B.
Incidence of anti-AZD9550 antibodies | Day 1 to Day 72
  • Incidence of ADA to AZD9550
  Applicable for Part B.
PD effect of AZD9550 on fasting glucose compared to placebo | From baseline to Week 24
  • Absolute change in fasting glucose
  Applicable for Parts C and D.
PD effect of AZD9550 on fasting lipid profile compared to placebo | From baseline to Week 24
  • Absolute and percentage change in total cholesterol, high-density lipoprotein, low-density lipoprotein, triglycerides, and BHB
  Applicable for Parts C and D.
The effect of AZD9550 on hepatic fat fraction versus placebo after 13 and 24 weeks of treatment | From baseline to Weeks 13 and 24
  * Change in hepatic fat fraction as measured by MRI-PDFF
  * Percent change in hepatic fat fraction as measured by MRI-PDFF
  Applicable for Part C.
Effects of AZD9550 compared to placebo on body weight | From baseline to Week 24
  * Change in body weight
  * Percent change in body weight • Proportion of participants achieving ≥ 5% body weight loss • Proportion of participants achieving ≥ 10% body weight loss
  * Absolute change in percentage body fat
  Applicable for Parts C and D.
Change in daily (24 hours) average glucose levels as measured by CGM | From baseline to Day 176
  Applicable for Parts C and D.
Change in fasting hepatic glycogen concentration adjusted for liver volume as measured by MRS | From baseline to Weeks 13 and 24
  Applicable for Part C.
Area Under concentration-time Curve of AZD9550 following repeat weekly SC doses | Day 1 to Day 169
  * AUC from 0 to the time of the last measured concentration (AUClast) at the first doses of each dose level and the last dose of MTD
  * AUC over a dosing interval (AUCtau) at the first doses of each dose level and the last dose of MTD
  Applicable for Parts C and D.
Incidence of anti-AZD9550 antibodies | Day 1 to Day 205
  • Incidence of ADA to AZD9550
  Applicable for Parts C and D.
Change in daily (24 hours) average glucose levels as measured by CGM | From baseline to Weeks 1, 2, 3, 4, 5, and 6, and during 14 days post last dose
  Applicable for Part A (excluding during 14 days post last dose). Applicable for Part B (excluding from baseline to Week 6 and during 14 days post last dose).
  Applicable for Parts C and D.
Change in 7-day average glucose levels as measured by CGM | From baseline to Weeks 1, 2, 3, 4, 5, and 6 and during 14 days post last dose
  Applicable for Part A (excluding during 14 days post last dose). Applicable for Part B (excluding from baseline to Week 6 and during 14 days post last dose).
  Applicable for Parts C and D.
Change in coefficient of variation of glucose levels as measured by CGM over 7 days | From baseline to Weeks 1, 2, 3, 4, 5, and 6, and during 14 days post last dose
  Applicable for Part A (excluding during 14 days post last dose). Applicable for Part B (excluding from baseline to Week 6 and during 14 days post last dose).
  Applicable for Parts C and D.
Change in percentage time spent in hyperglycaemia (> 140 mg/dL), normoglycaemia (70 -140 mg/dL), and clinically significant hypoglycaemia (< 54 mg/dL) as measured by CGM over 24 hours | From baseline to Weeks 1, 2, 3, 4, 5, and 6, and during 14 days post last dose
  Applicable for Part A (excluding during 14 days post last dose). Applicable for Part B (excluding from baseline to Week 6 and during 14 days post last dose).
  Applicable for Parts C and D.
Change in percentage time spent in hyperglycaemia (> 140 mg/dL), normoglycaemia (70 -140 mg/dL), and clinically significant hypoglycaemia (< 54 mg/dL) as measured by CGM over 7 days | From baseline to Weeks 1, 2, 3, 4, 5, and 6, and during 14 days post last dose
  Applicable for Part A (excluding during 14 days post last dose). Applicable for Part B (excluding from baseline to Week 6 and during 14 days post last dose).
  Applicable for Parts C and D.
Change in fasting hepatic glycogen concentration adjusted for liver volume as measured by MRS | From baseline to Week 5
  Applicable for Part B.
Percentage change in fasting hepatic glycogen concentration adjusted for liver volume as measured by MRS | From baseline to Week 5
  Applicable for Part B.
Change in fasting hepatic glycogen concentration unadjusted for liver volume as measured by MRS | From baseline to Week 5
  Applicable for Part B.
Percentage change in fasting hepatic glycogen concentration unadjusted for liver volume as measured by MRS | From baseline to Week 5
  Applicable for Part B.
Change in liver volume as measured by MRI | From baseline to Week 5
  Applicable for Part B.
Absolute change in body weight | From baseline to Week 5
  Applicable for Part B.
Percent change in body weight | From baseline to Week 5
  Applicable for Part B.
Proportion of participants achieving ≥ 5% body weight loss | From baseline to Week 5
  Applicable for Part B.
Proportion of participants achieving ≥ 10% body weight loss | From baseline to Week 5
  Applicable for Part B.
Change in 7-day average glucose levels as measured by CGM | From baseline to Day 176
  Applicable for Parts C and D.
Change in coefficient of variation of glucose levels as measured by CGM over 7 days | From baseline to Day 176 and during 14 days post last dose
  Applicable for Parts C and D.
Change in percentage time spent in hyperglycaemia (> 140 mg/dL), normoglycaemia (70 -140 mg/dL), and clinically significant hypoglycaemia (< 54 mg/dL) as measured by CGM over 24 hours | From baseline to Day 176
  Applicable for Parts C and D.
Change in percentage time spent in hyperglycaemia (> 140 mg/dL), normoglycaemia (70 -140 mg/dL), and clinically significant hypoglycaemia (< 54 mg/dL) as measured by CGM over 7 days | From baseline to Day 176 and during 14 days post last dose
  Applicable for Parts C and D.
Percentage change in fasting hepatic glycogen concentration adjusted for liver volume as measured by MRS | From baseline to Weeks 13 and 24
  Applicable for Part C.
Change in fasting hepatic glycogen concentration unadjusted for liver volume as measured by MRS | From baseline to Weeks 13 and 24
  Applicable for Part C.
Percentage change in fasting hepatic glycogen concentration unadjusted for liver volume as measured by MRS | From baseline to Weeks 13 and 24
  Applicable for Part C.
Change in liver volume, visceral and SC fat as measured by MRI | From baseline to Weeks 13 and 24
  Applicable for Part C.
Anti-AZD9550 antibody titre among participants with positive serum antibodies to AZD9550 | From Day 1 to 65
  • Titre of ADA to AZD9550
  Applicable for Part A.
Maximum observed concentration of AZD9550 following repeat weekly SC doses | Day to Day 72
  • Cmax at the last dose
  Applicable for Part B.
Half life associated with terminal phase elimination rate constant of AZD9550 following repeat weekly SC doses | Day 1 to Day 72
  • t1/2λz at the last dose
  Applicable for Part B.
Time to maximum observed concentration of AZD9550 following repeat weekly SC doses | Day 1 to Day 72
  • tmax at the last dose
  Applicable for Part B.
Apparent oral clearance of AZD9550 following repeat weekly SC doses | Day 1 to day 72
  • CL/F at the last dose
  Applicable for Part B.
Apparent volume of distribution of AZD9550 following repeat weekly SC doses | Day 1 to Day 72
  • Vz/F at the last dose
  Applicable for Part B.
Anti-AZD9550 antibody titre among participants with positive serum antibodies to AZD9550 | Day 1 to Day 72
  • Titre of ADA to AZD9550
  Applicable for Part B.
Maximum observed concentration of AZD9550 following repeat weekly SC doses | Day 1 to Day 169
  • Cmax at the first doses of each dose level and the last dose of MTD
  Applicable for Parts C and D.
Half life associated with terminal phase elimination rate constant of AZD9550 following repeat weekly SC doses | Day 1 to Day 169
  • t1/2λz at the first doses of each dose level and the last dose of MTD
  Applicable for Parts C and D.
Time to maximum observed concentration of AZD9550 following repeat weekly SC doses | Day 1 to Day 169
  • tmax at the first doses of each dose level and the last dose of MTD
  Applicable for Parts C and D.
Apparent oral clearance of AZD9550 following repeat weekly SC doses | Day 1 to Day 169
  • CL/F at the first doses of each dose level and the last dose of MTD
  Applicable for Parts C and D.
Apparent volume of distribution of AZD9550 following repeat weekly SC doses | Day 1 to day 169
  • Vz/F at the first doses of each dose level and the last dose of MTD
  Applicable for Parts C and D.
Anti-AZD9550 antibody titre among participants with positive serum antibodies to AZD9550 | Day 1 to Day 205
  • Titre of ADA to AZD9550
  Applicable for Parts C and D.
Change in visceral and subcutaneous fat as measured by MRI | From baseline to week 5
  Applicable for Part B.
PD effect of AZD9550 on glucose metabolism compared to placebo | From baseline to Week 4
  • Percent change in fasting glucose, fasting insulin, fasting c-peptide, and HbA1c
  Applicable for Part A.
PD effect of AZD9550 on glucose metabolism compared to placebo | From baseline to Week 5
  • Percent change in fasting glucose, fasting insulin, fasting c-peptide, and HbA1c
  Applicable for Part B.
PD effect of AZD9550 on glucose metabolism compared to placebo | From baseline to Week 24
  • Percent change in fasting glucose, fasting insulin, fasting c-peptide, and HbA1c
  Applicable for Parts C and D.
PD effect of AZD9550 on fasting insulin compared to placebo | From baseline to Week 4
  • Absolute change in fasting insulin
  Applicable for Part A.
PD effect of AZD9550 on fasting c-peptide compared to placebo | From baseline to Week 4
  • Absolute change in fasting c-peptide
  Applicable for Part A.
PD effect of AZD9550 on fasting insulin compared to placebo | From baseline to Week 24
  • Absolute change in fasting insulin
  Applicable for Parts C and D.
PD effect of AZD9550 on fasting c-peptide compared to placebo | From baseline to Week 24
  • Absolute change in fasting c-peptide
  Applicable for Parts C and D.
PD effect of AZD9550 on fasting insulin compared to placebo | From baseline to Week 5
  • Absolute change in fasting insulin
  Applicable for Part B.
PD effect of AZD9550 on fasting c-peptide compared to placebo | From baseline to Week 5
  • Absolute change in fasting c-peptide
  Applicable for Part B.
Absolute change in percentage body fat | From baseline to Week 5
  Applicable for Part B.
PD effect of AZD9550 on glucose metabolism following an MMTT compared to placebo | From baseline to Week 13 and Week 24
  * Percent change in glucose AUC(0-4h) measured by MMTT
  * Percent change in insulin AUC(0-4h) measured by MMTT
  * Percent change in c-peptide AUC(0-4h) measured by MMTT
  * Absolute change in fasting glucose, fasting insulin, and fasting c-peptide
  * Percent change in fasting glucose, fasting insulin, and fasting c-peptide
  Applicable for Part C.
PD effect of AZD9550 on HbA1c compared to placebo | From baseline to Week 4
  • Absolute change in HbA1c
  Applicable for Part A.
PD effect of AZD9550 on HbA1c compared to placebo | From baseline to Week 5
  • Absolute change in HbA1c
  Applicable for Part B.
PD effect of AZD9550 on HbA1c compared to placebo | From baseline to Week 24
  • Absolute change in HbA1c
  Applicable for Parts C and D.
Prevalence, incidence, and titres of ADAs to AZD9550 and AZD6234 in combination | After 24 weeks
  • To assess the immunogenicity profile of co-administered AZD9550 and AZD6234 in combination.
  Applicable for Part E.

CONTACTS AND LOCATIONS:
Locations (14):
- Austria (2):
  - Research Site, Graz
  - Research Site, Vienna
- Canada (5):
  - Research Site, Surrey, British Columbia
  - Research Site, Sarnia, Ontario
  - Research Site, Stouffville, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Sherbrooke, Quebec
- Germany (3):
  - Research Site, Magdeburg
  - Research Site, Neu-Ulm
  - Research Site, Neuss
- Japan (3):
  - Research Site, Fukuoka
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
- Research Site, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/